CLINICAL TRIAL: NCT01052857
Title: Efficacy of Acupuncture on Induction of Labor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Facchinetti Fabio, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: acupuncture
Record Dates: First submitted 2007-12-11; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2007-12

CONDITIONS: Labor; Pregnancy
Keywords: to evaluate acupuncture as possible alternative treatment for induction of labor; Induction; treatment; posterm
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): acupuncture daily fo 7 days
  Interventions: Procedure: acupuncture
- 2 (No Intervention): observation

INTERVENTIONS:
Procedure: acupuncture — acupuncture application
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of acupuncture for the induction of labor in pregnant women at the 40 weeks + 4 days of gestation.

DETAILED DESCRIPTION:
Women at 40+2-40+4 gestational age were allocated to receive acupuncture twice a week or observation in order to observe the efficacy of acupuncture in labour onset.

ELIGIBILITY:
Inclusion Criteria:

* Physiological pregnant women at 40 weeks + 4 days of gestation

Exclusion Criteria:

* Fetal or maternal disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the efficacy of acupuncture administered daily from 40 weeks + 4 days of gestation for induction of labor respect with placebo | 7 days

SECONDARY OUTCOMES:
to evaluate safety of acupuncture | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: facchinetti Fabio, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (2):
- Italy (2):
  - University of Modena and reggio emilia, Modena, modena
  - University of Modena and Reggio Emilia, Modena, Mo